CLINICAL TRIAL: NCT07074340
Title: Clinical Evaluation of Occlusal Stabilization Splints Fabricated Using Conventional Versus Fully Digital Workflow Based on Individual Mandibular Movements in TMD PATIENTS.
Brief Title: Clinical Evaluation of Occlusal Stabilization Splints Fabricated Using Conventional Versus Fully Digital Workflow
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mennatallah Mohamed Moustafa, assistant lecturer at Prosthodontics department, faculty of Dentistry,Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PROSR 3-3-12025
Record Dates: First submitted 2025-06-29; First posted 2025-07-20 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-05

CONDITIONS: Tempromandibular Joint Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Occlusal Splints manufactured with Conventional workflow (Active Comparator): maxillary and mandibular impressions will be made using rubber base impression material and the bite will be registered at centric by using rubber base bite registration material after patient deprogramming with Lucia jig. The occlusal record will be supplemented with a facebow transfer on a semi-adjustable articulator. The stabilization splint will be designed as wax-up then transferred to a duplicate cast for processing into heat-cured acrylic. After processing, the splint will be replaced on the master cast for occlusion refinement
  Interventions: Device: occlusal stabilization splint manufactured with a conventional workflow
- Occlusal Splints manufactured with fully-digital workflow (Experimental): For the intervention group; an intraoral scanner (Medit i700, South Korea) will be used to scan the maxillary and mandibular dentition and the maxillomandibular relationship in the centric relation position. A Jaw Tracking Device (JMA analyser; Zebris, Germany) will be used to record the jaw motion of the participants. The occlusal stabilization splints will be designed using a designing software (Exocad, USA). This device will be printed with a 3D printer (Creality, China) utilizing printable resin material.
  Interventions: Device: occlusal stabilization splint manufactured with Fully-digital workflow

INTERVENTIONS:
Device: occlusal stabilization splint manufactured with a conventional workflow — Heat-cured acrylic resin occlusal stabilization splint
  Arms: Occlusal Splints manufactured with Conventional workflow
Device: occlusal stabilization splint manufactured with Fully-digital workflow — 3D printed occlusal stabilization splints
  Arms: Occlusal Splints manufactured with fully-digital workflow

SUMMARY:
Temporomandibular disorders (TMDs) are considered one of the most common diseases in the dental clinic. TMDs are considered a major cause of chronic orofacial pain that affects the patient's daily activities and jaw function.

Occlusal splints are the most commonly used treatment modality for TMDs because of their low cost, ease of use and broad indications. Traditional workflow is complicated, technique sensitive and time-consuming as more chair-side time is required for occlusal adjustments . Recently, the revolutionary advances in digital technology have been widely used in prosthodontics, including the use of scanners, jaw tracking devices and CAD-CAM technologies. The fully digital workflow can offer more accuracy and less time consumption . However, literature is still limited and inconclusive regarding the use of fully digital workflows for occlusal splint construction.

DETAILED DESCRIPTION:
Stabilization splints (SS) are a major type of occlusal splints that is constructed from hard acrylic and designed to fully cover the maxillary and mandibular dentition in centric occlusion. They provide the patient with a stable occlusion in which the maximum number of simultaneous occlusal contacts, allows an adaptation of the TMJ apparatus and aids in self-repositioning of the condyle in the glenoid fossa.

Conventionally, the occlusal stabilization splint is made by fabrication a wax pattern on surveyed and mounted casts in centric relation then it is processed using lost wax technique to form a clear, heated-cured acrylic resin splint. The splints are thereafter tried intraorally and adjusted to obtain the desired adaptation to the teeth. The process of centric relation registration is complicated, technique sensitive and time- consuming. In addition, the conventional acrylic processing impairs the splint efficacy because of the presence of high porosity, high residual monomer content and shrinkage that affect the dimensional stability and accuracy.

Digital technology in prosthodontics has made revolutionary changes. The use of scanners, jaw tracking devices and CAD-CAM technologies has been involved widely regarding designing and manufacturing. This type of technology has demonstrated greater benefits in terms of dimensional stability, speed, better retention, and greater reproducibility. A study found that construction digitally printed stabilization splints with the use of intra-oral scanner and CAD-CAM showed the same patient improvement when compared to traditional workflow but with significant decrease in the required chairside time. Another concluded that the digital workflow was significantly preferred method among the participants during the construction of stabilization splints.

Recently, digital face bows and jaw tracking devices have been widely used used to record the mandibular movement and the jaw relationship for the fabrication of occlusal devices. These recent digital technologies can reduce the traditional errors and production time present in the conventional method of data acquisition for splints construction, which could improve the accuracy of occlusal splints and decrease the amount of intraoral occlusal adjustments that need to be made. There is a lack in the clinical trials investigating the use of jaw tracking device to acquire personalized articulator parameters to guide the production of occlusal stabilization splints. Hence, this clinical trial is aiming to compare chair side time and treatment outcomes (pain intensity and jaw functional limitation) of stabilization splints fabricated through a fully digital workflow using jaw tracking device for mandibular movement registration versus conventional workflow in patients with (TMDs).

ELIGIBILITY:
Inclusion criteria for participants:

* Age 20-40 years old.
* Complete dentition
* Intact and stable occlusion.
* TMD patients with more than one of following symptoms or signs: myofascial pain and /or pain in the TMJ, myofascial pain and/or pain in the TMJ on palpation, muscles tenderness, headache or earache

Exclusion criteria for participants:

* Patients with severe jaw functional limitations (jaw opening less than 3 fingers).
* Patients suffering from depression, anxiety or mental disorder.
* Patients with ongoing orthodontic treatments.
* History of a recent trauma to face, head or neck.
* Presence of dento-alveolar pathology.
* Presence of sever or moderate periodontitis.
* Patients with ongoing treatment related to TMD.

Exclusion Criteria:

-

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Chair side Time | "at record visit (baseline) and at delivery visit (during procedure)
  For both groups time lapsed during the records visit and fitting visit (T0) will be calculated with a stop watch.
  During the records visit, the time used for conventional and digital impressions, facebow record and jaw registration will be recorded in minutes. At fitting visit the necessary individual adjustments of the splints as well as, occlusion and articulation contact will be recorded in minutes.

SECONDARY OUTCOMES:
pain intensity | baseline and after 3 months
  Arabic translated instruments from the Axis II questionnaire form will be used to compare treatment outcome: Graded Chronic Pain Scale Version 2.0.

IPD SHARING:
Plan to Share IPD: No
security and privacy